CLINICAL TRIAL: NCT06616844
Title: Evaluating the Efficacy of Porcine Placental Extracellular Matrix Augmented Wound Care Against Standard Wound Care for the Management of Diabetic Foot Ulcers: A Multi-center, Prospective, Observer-blinded, Randomized Controlled Clinical Trial.
Brief Title: IDEAL: Efficacy of Porcine Placental Extracellular Matrix Augmented Plus Standard of Care (SOC) Versus SOC Alone for the Management of Diabetic Foot Ulcers
Acronym: IDEAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WC-24-453
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-03

CONDITIONS: Wound Heal; Ulcer
MeSH Terms: conditions — Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care (SOC) (No Intervention): Wound cleansing, using sterile saline, a non-ionic cleanser or a hypochlorous solution. Antiseptic agents including hydrogen peroxide, acetic acid, chlorhexidine, povidone/iodine, and cetrimide should not be used. Topical antimicrobials and silver dressings are also prohibited;
  Wound bed debridement, if clinically indicated.
  Primary wound dressings including a non-adherent, standard foam pad with or without a hydrogel beneath the dressing, or and alginate dressing, as is appropriate to maintain a moist wound environment while managing exudate;
  A secondary retention bandage appropriate to the amount of wound exudate, so as to avoid maceration of the peri-wound skin;
  Off-loading device appropriate to the location of wound with full length boot or total contact cast (unless not appropriate where a substitute off-loading device can be made with sponsor approval); and,
  Appropriate use of systemic antibiotics.
- Standard of Care + Intervention (Experimental): SOC arm with the following modifications:
  * Consecutive weekly application of PPECM for the 12-week study period.
  * Subjects will receive no more than 12 applications of PPECM
  Note: PPECM should be applied after standard wound cleansing and debridement procedures, prior to the application of primary wound dressing, in accordance with the IFU.
  Interventions: Device: InnovaMatrix® AC

INTERVENTIONS:
Device: InnovaMatrix® AC — SOC plus weekly application of the study device
  Other Names: Porcine Placental ExtraCellular Matrix (PPECM)
  Arms: Standard of Care + Intervention

SUMMARY:
A multi-center, prospective, observer-blinded, randomized controlled clinical trial to evaluate the efficacy of PPECM augmented standard of care versus standard of care alone in the management of hard-to-heal diabetic foot ulcers.

ELIGIBILITY:
Inclusion:

1. Subjects at least 21 years old. At least 50% of the enrolled population must be > 65 years of age.
2. Known history of type 1 or type 2 diabetes.
3. The patient must have a target ulcer meeting the following characteristics:

   i. A diabetic ulcer that is either Wagner Grade 1 or Wagner Grade 2 . ii. Located on the anatomical foot; defined as a minimum of 50% of ulcer area extending distal to the medial malleolus.

   iii. The target ulcer must have been present for a minimum of 4 weeks and no longer than 52 weeks.

   iv. The target ulcer must display evidence of delayed wound healing, defined as less than 50% wound area reduction over the four weeks preceding randomization.

   v. At randomization subjects must have a target ulcer with a minimum surface area of 1.0 cm2 and a maximum surface area of 25.0 cm2 measured post-debridement.
4. If two or more diabetic foot ulcers with the same Wagner Grade are present, the Index ulcer must additionally be:

   i. the ulcer with the largest wound area; ii. ≥ 2cm distant from any other ulcer on the affected limb, post-debridement; iii. the only ulcer to be evaluated by the study (one patient, one wound).
5. Subject has adequate circulation to the affected extremity, as demonstrated by at least one of the following within the past 30 days i. ABI ≥ 0.7 and ≤ 1.3; ii. TBI ≥ 0.6; iii. TCOM ≥ 40 mmHg; iv. PVR: biphasic.
6. BMI ≤45
7. Subject is willing to participate in all procedures and follow-up evaluations necessary to complete the study.
8. Subject has signed informed consent.

Exclusion:

1. The potential subject is known to have a life expectancy of <6 months.
2. Index Ulcers will be excluded if they meet any of the following criteria upon assessment:

   i. Index ulcer determined to be due to a condition other than diabetes ii. Active Charcot deformity OR major structural abnormalities of the foot iii. Known or suspected local skin malignancy to the index diabetic ulcer iv. Wound duration >12 months without intermittent closure
3. The target ulcer exhibits 2 or more of the following signs or symptoms consistent with clinical infection:

   i. erythema that extends ≥ 0.5cm from wound edge ii. local increased warmth iii. purulent exudate iv. local swelling or induration v. local tenderness or pain
4. Presence of osteomyelitis or exposed bone, probes to bone or joint capsule on investigator's exam or radiographic evidence.
5. The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent), radiation therapy, cytotoxic chemotherapy, or is taking medications that the Principal Investigator believes will interfere with wound healing (e.g., biologics).
6. The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
7. The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
8. The surface area of the target ulcer, as measured by digital planimetry or manual linear measurements (e.g. with a ruler), decreases by more than 25% in the 2 weeks prior to the initial screening visit ("historical" run-in period).
9. The surface area of the target ulcer, as measured by digital planimetry, decreases by more than 25% or more during the active 2-week screening phase: the 2 weeks from the initial screening visit (SV-1) to the TV-1 visit during which time the potential subject received SOC.
10. The potential subject is unable to adhere to therapeutic offloading, if required by anatomical location of target ulce.
11. Women who are pregnant or considering becoming pregnant within the next 6 months.
12. The potential subject has end stage renal disease requiring dialysis.
13. Participation in another clinical trial involving treatment with an investigational product within the previous 30 days.
14. A potential subject who, in the opinion of the Investigator, has a medical or psychological condition that may interfere with study assessments.
15. The potential subject was treated with hyperbaric oxygen therapy (HBOT) or a Cellular, Acellular, Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit.
16. The potential subject has a malnutrition indicator score <17 as measured on the Mini Nutritional Assessment.
17. Potential subjects with a sensitivity or allergy to porcine materials or collagen will be excluded.
18. Potential subjects with religious or personal objection to use of porcine- or animal-derived materials will be excluded.
19. A subject with a disorder that would create unacceptable risk of treatment complications is excluded.
20. Subjects will be considered ineligible for enrolment if any of the following criteria are met:

    i. Immune system disorders including Systemic Lupus Erythematosus (SLE), Acquired Immunodeficiency Syndrome (AIDS) or HIV.

    ii. In the past 6 months, having undergone a revascularization procedure aimed at increasing blood flow in the target limb OR any amputation affecting the target limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To determine if PPECM augmented care is superior to SOC in the closure of diabetic foot ulcers at 12 weeks. | 12 weeks
  Measure the incidence of complete wound closure, defined as 100% reepithelialization of the wound without drainage, confirmed at a second clinical visit occurring at least 2-weeks after the visit where wound closure was initially observed

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Angel City Research, Los Angeles, California
  - Center for Clinical Research, San Francisco, California
  - ILD Research Center, Vista, California
  - Dinamo Research and Diagnostic Center, Hialeah, Florida
  - Indiana Foot & Ankle, Jasper, Indiana
  - US-FAS, Hagerstown, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Northwell Health Comprehensive Wound Healing Center, New Hyde Park, New York
  - US-FAS, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No